CLINICAL TRIAL: NCT04458493
Title: Does Meal Replacement With a Carbohydrates and Protein Supplement Induce Weight Loss in Overweight and/or Obese Adults?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, Principal Investigator, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 116302
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Experimental): no supplement will be provided on the day of the experiment
  Interventions: Behavioral: satiety
- Generation UCAN (Experimental): carbohydrates - protein (Generation UCAN supplement, 400ml, 20% solution)
  Interventions: Behavioral: satiety; Dietary Supplement: Dietary Supplement: Generation UCAN supplementation

INTERVENTIONS:
Behavioral: satiety — satiety ratings, appetite and desire to eat (10-point visual analogue scale) will be measured at 30, 60 and 120 minutes after each meal replacement drink
Dietary Supplement: Dietary Supplement: Generation UCAN supplementation — meal replacement, Generation UCAN supplement, 400ml, 20% solution
  Arms: Generation UCAN

SUMMARY:
Participants will be randomized into two groups, one group will be the control (no intervention at all) and the other will be CHO-PRO (meal replacement, Generation UCAN supplement, 400ml, 20% solution). Prior to the start of the experiment, all participants will be asked to record their satiety ratings, appetite and desire to eat (10-point visual analogue scale) 30, 60 and 120 minutes after their regular dinner for 3 days. On the first day of the experiment, all participants will be asked to measure their waist and hip circumferences, fasting blood glucose level, maximal number of pushups and body weight using a scale at home prior to breakfast. Instructions on how to do the measurements properly will be recorded in a video and distributed to the participants. Participants in the control group will not receive any intervention. Participants in the CHO-PRO group will be provided with the supplement and they will be asked to consume the CHO - protein supplement (Generation UCAN supplement, 250ml, 10% solution) 6 to 7 hours after lunch, in place of their dinner for 6 weeks. They will also be asked to record their satiety ratings, appetite and desire to eat (10-point visual analogue scale) 30, 60 and 120 minutes after each meal replacement drink. All participants will be required to complete a dietary record, prior to, and during (at weeks 2 and 4) intervention. To track adherence of the CHO-PRO group, participants will be asked to check off the calendar that they did not consume the meal replacement due to various reasons. On day 43, all participants will be asked measure again waist and hip circumferences, fasting blood glucose level, maximal number of pushups and body weight using a scale at home prior to breakfast again.

ELIGIBILITY:
Inclusion Criteria:

* sedentary (<2 moderate exercise bouts/wk)
* between the ages of 18 to 40y
* body mass index (BMI) between >25

Exclusion Criteria:

* do not eat three meals a day typically
* taking medication that affects their eating patterns
* have metabolic and gastrointestinal diseases

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
changes in body weight | 1 day prior to the start of the experiment and on the 31st day of the experiment
  body weight will be measured using a scale at home prior to breakfast

SECONDARY OUTCOMES:
changes in waist and hip circumferences | 1 day prior to the start of the experiment and on the 31st day of the experiment
  waist and hip circumferences will be measured using a measuring tape at home prior to breakfast
changes in fasted blood glucose | 1 day prior to the start of the experiment and on the 31st day of the experiment
  blood glucose will be measured through finger pricks
changes in appetite ratings | 30, 60 and 120 minutes after each meal replacement drink
  appetite ratings will be asked with the use a 10 point visual analog scale (VAS), 10 being strong desire to consume food and 1 being no desire to consume food at all
changes in desire to eat ratings | 30, 60 and 120 minutes after each meal replacement drink
  desire to eat ratings will be asked with the use a 10 point visual analog scale (VAS), 10 being no desire to eat at all and 1 being strong desire to eat

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lemon, PhD, Principal Investigator — Western University

IPD SHARING:
Plan to Share IPD: No